CLINICAL TRIAL: NCT04738786
Title: Clinical Study Evaluating the Proper Surgical Safety Margin for Early Stage Oral Tongue Cancers: A Prospective Multicenter Randomized Non-inferiority Clinical Trial
Brief Title: Clinical Study Evaluating the Proper Surgical Safety Margin for Early Stage Oral Tongue Cancers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to Korean medical crisis, Resident strike, Patient referral (tongue cancer patients) to tertiary center has been in hold. Patient recruitment was seriously affected, and decreased.
Sponsor: Samsung Medical Center (Other)
Collaborators: Seoul National University Hospital (Other); Asan Medical Center (Other); Ajou University School of Medicine (Other); National Cancer Center, Korea (Other Government); Inje University (Other); Seoul National University Bundang Hospital (Other); Kangbuk Samsung Hospital (Other); Dong-A University Hospital (Other)
Responsible Party: Principal Investigator, Han-Sin Jeong, Director of Head and Neck Cancer Center, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-08-012
Record Dates: First submitted 2021-01-31; First posted 2021-02-04 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Tongue Cancer; Tongue Cancer TNM Staging Primary Tumor (T) T1; Tongue Cancer TNM Staging Primary Tumor (T) T2; Surgery; Resection Margin; Squamous Cell Carcinoma
Keywords: Tongue cancer; Surgery; Safety margin
MeSH Terms: conditions — Tongue Neoplasms; Margins of Excision; Carcinoma, Squamous Cell

STUDY DESIGN:
Intervention Model Description: A prospective multicenter randomized non-inferiority clinical trial, comparing two groups; 1.5 cm surgical safety margin versus 1.0 cm surgical safety margin in curative resection for cT1-2N0 oral tongue cancer
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Wide surgical safety margin (Active Comparator): 1.5 cm safety margin surgery for cT1-2N0 oral tongue cancer
  Interventions: Procedure: 1.5 cm surgical safety margin for cT1-2N0 oral tongue cancers
- Narrow surgical safety margin (Active Comparator): 1.0 cm safety margin surgery for cT1-2N0 oral tongue cancer
  Interventions: Procedure: 1.0 cm surgical safety margin for cT1-2N0 oral tongue cancers

INTERVENTIONS:
Procedure: 1.5 cm surgical safety margin for cT1-2N0 oral tongue cancers — Surgical resection including 1.5 cm normal tissue around the gross tumors
  Definition of safety margin: A surgical safety margin is defined as the margin of apparently non-tumorous tissue around a tumor that has been surgically removed (Resected normal-looking tissues from the gross tumor border). The surgical safety margin is applied to all directions of 3-dimensional tumors (mucosal and deep side).
  Arms: Wide surgical safety margin
Procedure: 1.0 cm surgical safety margin for cT1-2N0 oral tongue cancers — Surgical resection including 1.0 cm normal tissue around the gross tumors
  Arms: Narrow surgical safety margin

SUMMARY:
A prospective multicenter randomized non-inferiority clinical trial, to evaluate the efficacy and safety of 1.0 cm-safety margin surgery, compared with 1.5 cm safety margin surgery for cT1-2N0 oral tongue cancer

Summary:

A current standard primary treatment for oral tongue cancer is a curative surgical resection with/without adjuvant radiation treatments (or chemoradiation).

In pathological analysis of surgical specimens, more than 5 mm of non-tumorous tissues from the tumor border is regarded as a safe negative resection margin, according to the NCCN guideline (the National Comprehensive Cancer Network, Dec 10. 2020). To achieve this clear margin, surgeons are apt to use a 1.0 to 1.5 cm safety margin around the gross tumor during surgery, considering 30-50% tumor shrinkage in tissue fixation process.

Many previous retrospective data have been reported to suggest the optimal or proper surgical extent for oral tongue cancer. Wider resection can lead to better local control, however, it sacrifices more normal tissue, resulting in the functional deficit of tongue (speech and swallowing), even with reconstruction.

Unfortunately up to now, no prospective comparison of a different surgical safety margin for oral tongue cancer have been conducted to draw a more solid conclusion. Particularly in early stage oral tongue cancer (cT1-2N0), some study results have suggested that less than 5 mm resection margin in pathology specimens can be also safe and effective in terms of tumor control.

To achieve a well-grounded result about the proper surgical safety margin in early stage (cT1-2N0) oral tongue cancer, we will compare the outcomes of the two (1.5 cm versus 1.0 cm) surgical safety margin in curative resection for cT1-2N0 oral tongue cancer.

DETAILED DESCRIPTION:
Randomization

* The randomized allocation table was made by stratified block randomization methods with 1:1 ratio according to each participating surgeon and tumor stage.
* Baseline number (BN) should be provided to the subjects in the order of the date of surgery.

Surgical Procedure

* The study includes T1-2N0 oral tongue cancer patients. For the management of the primary lesion, wide resection with 1.0- or 1.5-cm surgical safety margin should be performed according to the results of study allocation.
* Neck management can be resection of primary tumor without neck dissection, with ipsilateral or bilateral neck dissection (guided by tumor location) or with sentinel lymph node biopsy, according to the NCCN guideline (version 1.2021).

Evaluation of the surgical safety margin

* The surgical safety margin should be meticulously evaluated in the pathology specimens in all directions.
* The surgical margins less than 0.3 or 0.5 cm in final pathology results are considered as the close surgical margin.

Adjuvant Treatment

* The adjuvant treatments either radiotherapy or chemoradiotherapy are conducted if indicated following the NCCN guideline.
* The follow-up after completion of the definitive treatment are made following the NCCN guideline.

Efficacy evaluation

* The primary outcomes are determined with 2-year local control rates after the completion of the curative treatments.
* The secondary outcomes are determined with the 5-year disease-free survival rates and speech/articulation functional analysis.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven oral tongue squamous cell carcinoma
* Stage cT1-2N0M0 tumors
* Treatment-naïve tumor
* American Society of Anesthesiologists (ASA) physical status classification 1-3.
* Patients who give a written informed consent voluntarily.

Exclusion Criteria:

* cT3-4 or N(+) tumors
* Recurrent tumors or salvage surgery
* Patients who have had a previous head and neck surgery and radiation treatment.
* Patients who have other head and neck cancer, within the last 5 years.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2021-01-18 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
2 year local control rate | 2 year
  At 2 years after the completion of treatment, % of local control (or recurrence rate)

SECONDARY OUTCOMES:
5 year recurrence free survival | 5 year
  5 year disease control rate
Speech function | 2 year
  Articulation score A seven-point articulation score (7: Within normal limits, 6 Mild-slight distortion and imprecision of consonants only, 5: Mild to moderate-all consonants targeted, 4: Moderate- at least 2 consonants placements acoustically distant from the target, 3: Moderate to marked-consonants and vowels both affected, 2: Marked- uses adaptive compensatory articulation for all lingual consonants, 1: Severe- does not use effective compensatory articulations) Reference: An objective assessment of speech and swallowing following free flap reconstruction for oral cavity cancers. Br J Plastic Surg 1996;49:363-9.
Swallowing function | 2 year
  Swallowing performance status score. A seven-point swallowing performance scale (1: Normal, 2: Within functional limits, 3: Mild impairment, 4, Mild-moderate, 5, Moderate, 6: Moderate-severe, 7: Severe impairment). (Reference: Swallowing Function in Patients With Head and Neck Cancer Prior to Treatment Arch Otolaryngol Head Neck Surg. 2000;126(3):371-377.)

CONTACTS AND LOCATIONS:
Overall Officials: Han-Sin Jeong, MD PhD, Principal Investigator — Head and Neck Cancer Center, Samsung Medical Center, Korea
Locations (4):
- South Korea (4):
  - Samsung Medical Center, Seoul
  - Asan Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Ajou university School of Medicine, Suwon

IPD SHARING:
Plan to Share IPD: No
The investigators will make our participant data available to other researchers after completion of this study.

REFERENCES:
- [Background] Jang JY, Choi N, Ko YH, Chung MK, Son YI, Baek CH, Baek KH, Jeong HS. Differential Impact of Close Surgical Margin on Local Recurrence According to Primary Tumor Size in Oral Squamous Cell Carcinoma. Ann Surg Oncol. 2017 Jun;24(6):1698-1706. doi: 10.1245/s10434-016-5497-4. Epub 2016 Aug 12. PMID 27519352